CLINICAL TRIAL: NCT06361017
Title: Research of the Prediction of Hemorrhage Transformation and Clinical Outcome by Cerebral Autoregulation After Endovascular Thrombectomy in Acute Ischemic Stroke Patients Caused by Middle Cerebral Artery or Internal Carotid Artery Occlusion.
Brief Title: The Prediction of Hemorrhage Transformation by Cerebral Autoregulation in AIS Patient After Endovascular Thrombectomy
Acronym: PHASE
Status: Enrolling by invitation | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: QNPY2022007
Record Dates: First submitted 2024-03-26; First posted 2024-04-11 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-04

CONDITIONS: Acute Ischemic Stroke; Endovascular Thrombectomy; Dynamic Cerebral Autoregulation
Keywords: Acute Ischemic Stroke; ultrasound; endovascular thrombectomy; dynamic cerebral autoregulation; Hemodynamics
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- favorable outcome group: The favorable outcome group was defined as the modified Rankin Scale (mRS) score ≤2 in the AIS patients at 3 months after endovascular thrombectomy.
  Interventions: Procedure: endovascular thrombectomy
- unfavorable outcome group: The unfavorable outcome group was defined as the modified Rankin Scale (mRS) score with 3-6 in the AIS patients at 3 months after endovascular thrombectomy.
  Interventions: Procedure: endovascular thrombectomy
- HT group: HT group was defined as the AIS patients have hemorrhage transformation in 7 days after endovascular thrombectomy.
  Interventions: Procedure: endovascular thrombectomy
- non-HT group: Non-HT group was defined as the AIS patients do not have hemorrhage transformation in 7 days after endovascular thrombectomy.
  Interventions: Procedure: endovascular thrombectomy

INTERVENTIONS:
Procedure: endovascular thrombectomy — All individuals were anesthetized, with local or general anesthesia dependent on the cooperation level of the patient. During the procedure, it was mandatory to administer intravenous heparin to maintain the activated clotting time between 250 and 300 s, except for subjects who received intravenous alteplase. The procedures were performed through the femoral artery. The selection of stent retriever type and size, along with any required devices, such as guide wires and catheters, as well as the intervention strategy, was at the interventionists' discretion.
  Other Names: mechanical thrombectomy

SUMMARY:
This observational study was designed for observe the cerebral hemodynamics and dynamic cerebral autoregulation (dCA) after endovascular thrombectomy (EVT) in acute ischemic stroke (AIS) patients. And analysis the relationship between the dCA damage degree and hemorrhage transformation (HT) and clinical outcome.

Patients: patients with AIS caused by middle cerebral artery or internal carotid artery occlusion who accepted EVT.

dCA Examination: dCA examinations were performed at 24 hours, 48 hours, 72 hours, and 5 days after EVT.

The objectives of the study were as follows: The changes of cerebral hemodynamics and parameters of dCA in different time periods after EVT were analyzed. So as to determine the correlation between hemodynamics and dCA change and HT and clinical outcome after EVT and to explore the predictors of HT and adverse clinical outcomes.

DETAILED DESCRIPTION:
Part of the data from March 2022 to March 2022 was obtained, but it was still need more data and need a one-year follow-up of the data. Therefore, this is a 4 years prospective cohort study.

The objectives of the study were as follows: This observational study was designed for observe the cerebral hemodynamics and dynamic cerebral autoregulation (dCA) after endovascular thrombectomy (EVT) in acute ischemic stroke (AIS) patients. And analysis the relationship between the dCA damage degree and hemorrhage transformation (HT) and clinical outcomes. To explore the predictors of HT and adverse clinical outcomes.

A. To enroll 300 cases of patients with AIS caused by middle cerebral artery or internal carotid artery occlusion who accepted EVT.

B. dCA examinations were performed at 24 hours, 48 hours, 72 hours, and 5 days after EVT.

C. The computed tomography was performed to distinguish if the patients have HT within 7 days after EVT.

D. Utilizing the modified Rankin Scale (mRS), the clinical prognosis was assessed 3 months and 1 year after stroke. The outcomes were dichotomized according to the mRS score: favorable outcome (mRS ≤ 2) and unfavorable outcome (mRS: 3-6). During the telephone call follow-up, the clinician was unaware of any pertinent clinical or dCA information while examining each mRS score.

E. All tests are non-invasive.

ELIGIBILITY:
Inclusion Criteria:

* (i) age ≥18 years; (ii) complete recanalization of the affected MCA (thrombolysis in cerebral infarction grade 2b or 3); and (iii) sufficient temporal windows to obtain ﬂow signals for the MCA.

Exclusion Criteria:

* (i) inability to perform dCA after EVT due to restlessness; (ii) re-occlusion of the culprit MCA after EVT; and (iii) other conditions such as low cerebral blood ﬂow caused by severe heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients 18 years of age and older with acute ischemic stroke who underwent endovascular thrombectomy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence of hemorrhage transformation | 7 days
  The AIS patients have hemorrhage transformation detected by head computed tomography scans within 7 days after EVT
Patients without hemorrhage transformation | 7 days
  The AIS patients do not have hemorrhage transformation detected by head computed tomography scans within 7 days after EVT
The occurrence of unfavorable outcome | 3 months
  The modified Rankin Scale (mRS) score was 3-6 of AIS patients with EVT after 3 months.
The occurrence of favorable outcome | 3 months
  The modified Rankin Scale (mRS) score ≤2 of AIS patients with EVT after 3 months.

SECONDARY OUTCOMES:
The occurrence of long-term unfavorable outcome | 1 year
  The modified Rankin Scale (mRS) score was 3-6 of AIS patients with EVT after 1 year.
The occurrence of long-term favorable outcome | 1 year
  The modified Rankin Scale (mRS) score ≤2 of AIS patients with EVT after 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Yingqi Xing, M.D., Principal Investigator — Department of Vascular Ultrasonography, Xuanwu Hospital.
Locations (1):
- Department of Vascular Ultrasonography, Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tian G, Ji Z, Huang K, Lin Z, Pan S, Wu Y. Dynamic cerebral autoregulation is an independent outcome predictor of acute ischemic stroke after endovascular therapy. BMC Neurol. 2020 May 15;20(1):189. doi: 10.1186/s12883-020-01737-w. PMID 32414382
- [Background] Nogueira RG, Jadhav AP, Haussen DC, Bonafe A, Budzik RF, Bhuva P, Yavagal DR, Ribo M, Cognard C, Hanel RA, Sila CA, Hassan AE, Millan M, Levy EI, Mitchell P, Chen M, English JD, Shah QA, Silver FL, Pereira VM, Mehta BP, Baxter BW, Abraham MG, Cardona P, Veznedaroglu E, Hellinger FR, Feng L, Kirmani JF, Lopes DK, Jankowitz BT, Frankel MR, Costalat V, Vora NA, Yoo AJ, Malik AM, Furlan AJ, Rubiera M, Aghaebrahim A, Olivot JM, Tekle WG, Shields R, Graves T, Lewis RJ, Smith WS, Liebeskind DS, Saver JL, Jovin TG; DAWN Trial Investigators. Thrombectomy 6 to 24 Hours after Stroke with a Mismatch between Deficit and Infarct. N Engl J Med. 2018 Jan 4;378(1):11-21. doi: 10.1056/NEJMoa1706442. Epub 2017 Nov 11. PMID 29129157
- [Result] Zhao W, Liu R, Yu W, Wu L, Wu C, Li C, Li S, Chen J, Song H, Hua Y, Ma Q, Ji X. Elevated pulsatility index is associated with poor functional outcome in stroke patients treated with thrombectomy: A retrospective cohort study. CNS Neurosci Ther. 2022 Oct;28(10):1568-1575. doi: 10.1111/cns.13888. Epub 2022 Jun 16. PMID 35707901